CLINICAL TRIAL: NCT06364449
Title: Clinical Decision Tree Analysis of Hemodialysis Arteriovenous Access Choices and Creations - a Multiple-center Retrospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Assistant professor, National Taiwan University Hospital
Other Study IDs: 202309052RIND
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Decision Tree Analysis
Keywords: Arteriovenous Fistula; AV graft; Hemodialysis; decision tree analysis
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- AVF-wrist
  Interventions: Other: No intervention
- AVF-elbow
  Interventions: Other: No intervention
- AVG-forearm
  Interventions: Other: No intervention
- AVG-elbow
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Our study aim was to utilize a decision tree analysis (DTA) model to gain insight into the decision-making process within a multiple-center cohort.

DETAILED DESCRIPTION:
Scientific research focuses on limited parameters, aims to confirm hypotheses, and has minor uncertainties. In contrast, medical decisions involve many unknowns. Physicians must use all available knowledge to make the best decisions. However, decision-making can become unpredictable when limited evidence exists, leading to non-reproducible outcomes.

According to clinical guidelines, patients who need pre-kidney replacement therapy (pre-KRT) and opt for hemodialysis (HD) with a reasonable life expectancy should have arteriovenous (AV) access created. Nevertheless, constructing an AVF has limitations. [Additionally, the maturation rate of AVF is suboptimal. Therefore, after careful consideration of the patient's end-stage kidney disease (ESKD) life plan, the suggested order of AV access types and locations starts a native distal forearm radiocephalic AVF, followed by a native proximal forearm AVF, a forearm arteriovenous graft (AVG), then an upper arm AVG creation.[Lok et al., 2020] However, the decision-making process for selecting hemodialysis access is shared between patients, physicians, and the surgeon's discretion.

Therefore, clinical kidney practice requires effective decision-making to address ESKD life plan and AV access concerns while minimizing harm. Decision analysis models can bridge the gap between research and decision-making. Our study aim was to utilize a decision tree analysis (DTA) model to gain insight into the decision-making process within a multiple-center cohort.

ELIGIBILITY:
Inclusion Criteria:

- adult patients between the ages of 18 and 80 who were referred for primary hemodialysis (HD) AV access creation. We included those in the pre-kidney replacement therapy (pre-KRT) stage and those who in the early end-stage kidney disease (ESKD) urgently started HD without sufficient time to plan for AV access

Exclusion Criteria:

- patients who underwent a secondary AV access surgery, like a transposed radiobasilic AVF or a revision of AVG.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic kidney disease (CKD) and were in the pre-kidney replacement therapy (pre-KRT) stage, requiring their first hemodialysis (HD) AV access creatio
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
predicted AV access choices | postoperativ 3 -12 months
  identifying parameters that predicted AV access choices among the four types

SECONDARY OUTCOMES:
to determine factors affecting clinical use of the targeted AV access over a variable timeframe | postoperativ 3 -12 months
  The secondary objective was to determine factors affecting clinical use of the targeted AV access over a variable timeframe

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yang Chan, phd, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan